CLINICAL TRIAL: NCT02913261
Title: A Phase III Randomized Open-label Multi-center Study of Ruxolitinib Versus Best Available Therapy in Patients With Corticosteroid-refractory Acute Graft vs. Host Disease After Allogeneic Stem Cell Transplantation
Brief Title: Safety and Efficacy of Ruxolitinib Versus Best Available Therapy in Patients With Corticosteroid-refractory Acute Graft vs. Host Disease After Allogeneic Stem Cell Transplantation
Acronym: REACH2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC424C2301; 2016-002584-33 (EudraCT Number)
Record Dates: First submitted 2016-09-18; First posted 2016-09-23 (Estimated); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-05

CONDITIONS: Corticosteroid Refractory Acute Graft vs Host Disease
Keywords: GvHD (Graft versus Host Disease); INC424; ruxolitinib; best available therapy (BAT); corticosteroid-refractory acute graft vs. host disease; allogeneic stem cell transplantation; steroid refractory acute graft vs. host disease; Janus Kinase (JAK) inhibitor
MeSH Terms: conditions — Graft vs Host Disease | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib (Experimental): These patients were administered Ruxolitinib orally twice per day (b.i.d) at a dose of 10 mg bid, as two 5-mg tablets. Ruxolitinib was taken without regards to food.
  Interventions: Drug: Ruxolitinib (RUX)
- Best Available Therapy (BAT) (Active Comparator): These patients were administered BAT per the Investigator's best judgement based on a specific list of BAT.
  Interventions: Drug: Best Available Therapy (BAT)

INTERVENTIONS:
Drug: Ruxolitinib (RUX) — Ruxolitinib was provided as 5 mg tablets for oral use.
  Other Names: INC424
  Arms: Ruxolitinib
Drug: Best Available Therapy (BAT) — BAT was based on the investigator's best judgment, taking into account the manufacturer's instructions, labeling, patient's medical condition, and institutional guidelines for any dose adjustment. The BAT in this study was identified by the investigator prior to patient randomization among the following treatments currently used in this setting: anti-thymocyte globulin (ATG), extracorporeal photopheresis (ECP), mesenchymal stromal cells (MSC), low-dose methotrexate (MTX), mycophenolate mofetil (MMF), mTOR inhibitors (everolimus or sirolimus), etanercept, or infliximab. No other types or combinations of BAT were permitted.
  Arms: Best Available Therapy (BAT)

SUMMARY:
Assess the efficacy and safety of ruxolitinib compared to Best Available Therapy (BAT) in patients with corticosteroid-refractory acute graft vs. host disease (aGvHD) after allogeneic stem cell transplantation.

DETAILED DESCRIPTION:
This randomized, phase III, open-label study investigated the efficacy and safety of ruxolitinib vs. BAT added to the patient's immunosuppressive regimen in adults and adolescents (≥ 12 years old) with grade II-IV Steroid-refractory Acute Graft vs. Host Disease (SR-aGvHD). During the screening period, patients were monitored for a diagnosis of SR-aGvHD, which was defined as patients who had high-dose systemic corticosteroids (methylprednisolone 2 mg/kg/day [or equivalent prednisone dose 2.5 mg/kg/day]), given alone or combined with CNI, who either:

1. Progressed based on organ assessment after at least 3 days compared to organ stage at the time of initiation of high-dose systemic corticosteroid +/- CNI for the treatment of Grade II-IV aGvHD, OR
2. Failed to achieve at a minimum a partial response based on organ assessment after 7 days compared to organ stage at the time of initiation of high-dose systemic corticosteroid +/- CNI for the treatment of Grade II-IV aGvHD, OR
3. Failed corticosteroid taper defined as fulfilling either one of the following criteria:

   * Requirement for an increase in the corticosteroid dose to methylprednisolone ≥ 2 mg/kg/day (or equivalent prednisone dose ≥ 2.5 mg/kg/day) OR
   * Failure to taper the methylprednisolone dose to <0.5 mg/kg/day (or equivalent prednisone dose <0.6 mg/kg/day) for a minimum 7 days.

Patients meeting eligibility criteria were randomized 1:1 to receive either ruxolitinib or BAT stratifying on aGvHD grade at the time of randomization (Grade II vs III vs IV).

Study treatment began on Day 1 (no later than 72 hours after randomization) followed by regular visits for assessments of efficacy and safety. Study treatment was administered until the patient met any of the criteria for discontinuation of study treatment or, in responders (i.e. patients achieving PR or CR) until the dosing schedule for ruxolitinib or BAT was completed.

All responders were to be tapered off during the treatment period by, first tapering from corticosteroids, followed by CNI and ruxolitinib. A slow tapering extending beyond 24 weeks was permitted for ruxolitinib at Investigator's discretion rather than an abrupt cessation, as the latter could result in an aGvHD flare.

During the Treatment Period, patients randomized to BAT could have crossed over to ruxolitinib between Day 28 and Week 24 if they:

* Failed to meet the primary endpoint response definition (CR or PR) at Day 28 OR
* Lost the response thereafter and met criteria for progression, mixed response, or no response, necessitating new additional systemic immunosuppressive treatment for aGvHD.

AND

- Did not have signs/symptoms of chronic Graft vs. Host Disease (cGvHD) (overlap syndrome, progressive, or de novo cGvHD)

Patients who crossed over to ruxolitinib were followed until completion of treatment with ruxolitinib and received the same treatment and tapering schedule as patients randomized to ruxolitinib treatment.

The End of Treatment (EOT) visit occurred when the patient completed the study treatment period or earlier if the patient met any of the criteria for discontinuation of study treatment.

Patient's treatment period was up to 6 months (Week 24). However, ruxolitinib taper could be delayed up to 2 years from randomization due to an aGvHD flare or other safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone Allogeneic Stem Cell Transplanttaion (alloSCT) from any donor source (matched unrelated donor, sibling, haplo-identical) using bone marrow, peripheral blood stem cells, or cord blood. Recipients of non- myeloablative, myeloablative, and reduced intensity conditioning are eligible
* Clinically diagnosed Grades II to IV acute GvHD as per standard criteria occurring after alloSCT requiring systemic immune suppressive therapy. Biopsy of involved organs with aGvHD is encouraged but not required for study screening.
* Confirmed diagnosis of steroid refractory aGvHD defined as patients administered high-dose systemic corticosteroids (methylprednisolone 2 mg/kg/day [or equivalent prednisone dose 2.5 mg/kg/day]), given alone or combined with calcineurin inhibitors (CNI) and either:

  * Progressing based on organ assessment after at least 3 days compared to organ stage at the time of initiation of high-dose systemic corticosteroid +/- CNI for the treatment of Grade II-IV aGvHD, OR
  * Failure to achieve at a minimum partial response based on organ assessment after 7 days compared to organ stage at the time of initiation of high-dose systemic corticosteroid +/- CNI for the treatment of Grade II-IV aGvHD,OR
  * Patients who fail corticosteroid taper defined as fulfilling either one of the following criteria:
* Requirement for an increase in the corticosteroid dose to methylprednisolone ≥2 mg/kg/day (or equivalent prednisone dose ≥2.5 mg/kg/day) , OR
* Failure to taper the methylprednisolone dose to <0.5 mg/kg/day (or equivalent prednisone dose <0.6 mg/kg/day) for a minimum 7 days.

Exclusion Criteria:

* Has received more than one systemic treatment for steroid refractory aGvHD.
* Presence of an active uncontrolled infection including significant bacterial, fungal, viral or parasitic infection requiring treatment. Infections are considered controlled if appropriate therapy has been instituted and, at the time of screening, no signs of progression are present. Progression of infection is defined as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Evidence of uncontrolled viral infection including Cytomegalovirus (CMV), Epstein-Barr Virus (EBV), Human Herpes Virus-6 (HHV-6), Hepatitis Virus (HBV), or Hepatitis C Virus (HCV) based on assessment by the treating physician.
* Presence of relapsed primary malignancy, or who have been treated for relapse after the alloHSCT was performed, or who may require rapid immune suppression withdrawal as pre-emergent treatment of early malignancy relapse.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2021-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (92):
- Australia (4):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Linz
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (7):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Saskatoon, Saskatchewan
- Novartis Investigative Site, Prague, Czech Republic, Czechia
- Novartis Investigative Site, Copenhagen, Denmark
- France (12):
  - Novartis Investigative Site, Saint Priest En Jarez, Pays de la Loire Region
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (15):
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Thessaloniki, GR, Greece
- Novartis Investigative Site, Hong Kong, Hong Kong
- Israel (4):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Tel Aviv
- Italy (11):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, San Giovanni Rotondo, FG
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Udine, UD
- Japan (14):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Minato Ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Utrecht, The Netherlands, Netherlands
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Seoul, South Korea
- Spain (7):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Taichung, Taiwan
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- United Kingdom (2):
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mohty M, Socie G, Szer J, Niederwieser D, Butler J, Wagner-Drouet E, Or R, Rovenvald-Zuckerman T, Bozdag SC, Forcade E, Grillo G, Kroger N, Stolzel F, Russo D, Sanz J, Sarkar R, Stefanelli T, Wilke C, Zeiser R, von Bubnoff N. Ruxolitinib Versus Best Available Therapy in Patients With Steroid-Refractory Acute Graft-Versus-Host Disease: Final Analysis From the Randomized Phase III REACH2 Trial. J Clin Oncol. 2025 Dec;43(34):3639-3645. doi: 10.1200/JCO-25-00809. Epub 2025 Oct 15. PMID 41092247
- [Derived] Mahmoudjafari Z, Kintsch E, Xue Z, Bhatt V, Galvin J, Locatelli F, Zeiser R. Impact of concomitant azoles on ruxolitinib treatment in patients with GVHD: post hoc analyses of REACH2 and REACH3. Blood Adv. 2025 Aug 26;9(16):4206-4216. doi: 10.1182/bloodadvances.2025016212. PMID 40472328
- [Derived] Socie G, Niederwieser D, von Bubnoff N, Mohty M, Szer J, Or R, Garrett J, Prahallad A, Wilke C, Zeiser R. Prognostic value of blood biomarkers in steroid-refractory or steroid-dependent acute graft-versus-host disease: a REACH2 analysis. Blood. 2023 Jun 1;141(22):2771-2779. doi: 10.1182/blood.2022018579. PMID 36827620
- [Derived] Zeiser R, von Bubnoff N, Butler J, Mohty M, Niederwieser D, Or R, Szer J, Wagner EM, Zuckerman T, Mahuzier B, Xu J, Wilke C, Gandhi KK, Socie G; REACH2 Trial Group. Ruxolitinib for Glucocorticoid-Refractory Acute Graft-versus-Host Disease. N Engl J Med. 2020 May 7;382(19):1800-1810. doi: 10.1056/NEJMoa1917635. Epub 2020 Apr 22. PMID 32320566
- [Derived] Jagasia M, Zeiser R, Arbushites M, Delaite P, Gadbaw B, Bubnoff NV. Ruxolitinib for the treatment of patients with steroid-refractory GVHD: an introduction to the REACH trials. Immunotherapy. 2018 Apr;10(5):391-402. doi: 10.2217/imt-2017-0156. Epub 2018 Jan 10. PMID 29316837

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 310 patients with SR-aGvHD were enrolled, out of which 309 patients were included in the analysis (as one patient did not sign the study informed consent prior to receiving BAT (protocol deviation) and was excluded from all analyses).
  Completed = Completed the treatment period Not completed = Discontinued from treatment period
Pre-assignment Details: The screening period ranged from Day -28 to Day -1. Screening activities and assessment of inclusion and exclusion criteria began once the patient was diagnosed with aGvHD. Any occurrence of SR-aGvHD was monitored closely.
Groups:
- Ruxolitinib (RUX): These patients were administered Ruxolitinib orally twice per day (b.i.d) at a dose of 10 mg bid, as two 5-mg tablets. Ruxolitinib was taken without regards to food.
Period: Overall Study
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Started | 154 | 155
Not Treated | 2 | 5
Crossover Treatment at End of Randomized Treatment | 0 | 49
Entered Long-term Follow-up | 102 | 51
Completed Screening & Randomized | 154 | 155
Completed Screening & Not Randomized | 0 | 1
Completed (Completed = Completed the treatment period Not Completed = Discontinued from treatment period) | 35 | 20
Not Completed | 119 | 135
Not completed — Technical problems | 0 | 1
Not completed — Lack of Efficacy | 32 | 69
Not completed — Adverse Event | 27 | 5
Not completed — Death | 25 | 22
Not completed — Failure to meet protocol continuation criteria | 13 | 10
Not completed — Disease relapse | 8 | 13
Not completed — Physician Decision | 8 | 9
Not completed — Subject/guardian decision | 4 | 6
Not completed — Graft loss | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT) | Total
Number analyzed (Participants) | 154 | 155 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (16.30) | 50.9 (14.97) | 49.5 (15.69)
Age, Customized [Number; unit: Participants]
  Adolescents, 12 - <18 years | 5 | 4 | 9
  18 - 65 years | 128 | 126 | 254
  >65 years | 21 | 25 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 64 | 126
  Male | 92 | 91 | 183
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 111 | 102 | 213
  Black or African American | 0 | 1 | 1
  Asian | 19 | 29 | 48
  Other | 8 | 4 | 12
  Unknown | 16 | 19 | 35
Weight [Mean (Standard Deviation); unit: kg] — Population: the weight at baseline was missing for 7 patients
  kg
    number analyzed (Participants) | 150 | 152 | 302
    (all) | 67.5 (14.04) | 66.2 (14.78) | 66.9 (14.41)

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) at Day 28
Description: Overall response rate at Day 28 after randomization was defined as the percentage participants in each arm demonstrating a complete response (CR) or partial response (PR), based on investigator assessment & according to standard criteria, without requirement for additional systemic therapies for an earlier progression, mixed response or non-response. Scoring of response was relative to the organ stage at the time of randomization.
  CR was defined as a score of 0 for the aGvHD grading in all evaluable organs that indicates complete resolution of all signs & symptoms of aGvHD in all evaluable organs without administration of additional systemic therapies for any earlier progression, mixed response or non-response of aGvHD.
  PR was defined as improvement of 1 stage in 1 or more organs involved with aGvHD signs or symptoms without progression in other organs or sites without administration of additional systemic therapies for an earlier progression, mixed response or non-response of aGvHD.
Time Frame: Day 28
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 154 | 155
Percentage of participants | 62.3 [54.2 to 70.0] | 39.4 [31.6 to 47.5]
Statistical Analysis 1: Comparison: Ruxolitinib (RUX) vs Best Available Therapy (BAT); Test type: Superiority; p < .0001, Stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.64, 95% CI 2-sided [1.65 to 4.22]

2. Secondary Outcome: Durable Overall Response Rate (DORR) (Key Secondary Endpoint) at Day 56
Description: Percentage of all participants in each arm who achieved a complete response (CR) or partial response (PR) at Day 28 (primary endpoint) AND maintained a CR or PR at Day 56 based on investigator assessment and according to standard criteria.
  CR was defined as a score of 0 for the aGvHD grading in all evaluable organs that indicates complete resolution of all signs and symptoms of aGvHD in all evaluable organs without administration of additional systemic therapies for any earlier progression, mixed response or non-response of aGvHD.
  PR was defined as improvement of 1 stage in 1 or more organs involved with aGvHD signs or symptoms without progression in other organs or sites without administration of additional systemic therapies for an earlier progression, mixed response or non-response of aGvHD.
Time Frame: Day 56
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 154 | 155
Percentage of participants | 39.6 [31.8 to 47.8] | 21.9 [15.7 to 29.3]
Statistical Analysis 1: Comparison: Ruxolitinib (RUX) vs Best Available Therapy (BAT); Test type: Superiority; p = 0.0005, Stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.38, 95% CI 2-sided [1.43 to 3.94]

3. Secondary Outcome: Overall Response Rate (ORR) at Day 14
Description: ORR at Da4 14 is the percentage of participants who achieved overall response (CR+PR) at Day 14 based on investigator assessment and according to standard criteria.
  CR was defined as a score of 0 for the aGvHD grading in all evaluable organs that indicates complete resolution of all signs and symptoms of aGvHD in all evaluable organs without administration of additional systemic therapies for any earlier progression, mixed response or non-response of aGvHD.
  PR was defined as improvement of 1 stage in 1 or more organs involved with aGvHD signs or symptoms without progression in other organs or sites without administration of additional systemic therapies for an earlier progression, mixed response or non-response of aGvHD.
Time Frame: Day 14
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 154 | 155
Percentage of participants | 63.0 [54.8 to 70.6] | 47.1 [39.0 to 55.3]
Statistical Analysis 1: Comparison: Ruxolitinib (RUX) vs Best Available Therapy (BAT); Test type: Superiority; p = 0.0029, Stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.98, 95% CI 2-sided [1.24 to 3.17]

4. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was defined for patients who had a CR or PR at Day 28. This was the interval between the date of first documented response of CR or PR (i.e., the start date of response), till the date of progression or addition of systemic therapies for aGvHD on or after Day 28. Death without prior observation of aGvHD progression and onset of chronic GvHD were considered. Duration of response was censored at the last response assessment prior to or at the analysis cut-off date, if no events/competing risk occurred before or at the cut-off date.
Time Frame: Up to 24 months
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization. These were patients to whom study treatment was assigned by randomization and whose overall response was complete response (CR) or partial response (PR).
Measure: Median (Full Range); unit: Days
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 98 | 62
Days | 167.0 [22.0 to 677.0] | 106.0 [10.0 to 526.0]

5. Secondary Outcome: Cumulative Steroid Dosing Until Day 56
Description: Weekly cumulative steroid dose for each participant up to Day 56 or discontinuation of randomized treatment. Participants should have undergone tapering of steroids if it had been required. Tapering the immunosuppression therapy was performed in 2 steps: Taper of corticosteroids: initiated not earlier than Day 7, and performed as per institutional guidelines. Only patients with assessments done at each time point are reported. This is the reason that the overall number per treatment is higher and the number of participants with responses vary over time.
Time Frame: up to Day 56
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Median (Full Range); unit: mg
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 154 | 155
mg
  By Week 1: number analyzed (Participants) | 151 | 154
  By Week 1 | 962.5 [140.0 to 2337.5] | 923.6 [140.0 to 6093.8]
  By Week 2: number analyzed (Participants) | 150 | 150
  By Week 2 | 1740.0 [280.0 to 3500.0] | 1725.0 [280.0 to 7173.3]
  By Week 3: number analyzed (Participants) | 143 | 141
  By Week 3 | 2375.0 [350.0 to 5250.0] | 2340.0 [370.0 to 8000.0]
  By Week 4: number analyzed (Participants) | 132 | 136
  By Week 4 | 2866.9 [420.0 to 7000.0] | 2816.3 [420.0 to 9050.0]
  By Week 5: number analyzed (Participants) | 124 | 106
  By Week 5 | 3268.1 [455.0 to 8750.0] | 3290.6 [420.0 to 9825.0]
  By Week 6: number analyzed (Participants) | 115 | 84
  By Week 6 | 3606.3 [490.0 to 10500.0] | 3543.8 [420.0 to 10435.0]
  By Week 7: number analyzed (Participants) | 107 | 75
  By Week 7 | 3850.0 [495.0 to 11250.0] | 3706.3 [420.0 to 10955.0]
  By Week 8: number analyzed (Participants) | 87 | 67
  By Week 8 | 4000.0 [857.5 to 9475.0] | 4006.3 [420.0 to 11875.0]

6. Secondary Outcome: Kaplan Meier Estimates of Probability of Overall Survival (OS) by Time Interval
Description: OS was defined as the time from the date of randomization to date of death due to any cause. If a patient was not known to have died, then OS was censored at the latest date the patient was known to be alive (on or before the cut-off date). Results are based on Kaplan Meier (KM) estimates.
Time Frame: 1, 2, 6, 12, 18 & 24 months
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 154 | 155
Percentage of participants
  1 Month | 90.04 [84.02 to 93.87] | 85.48 [78.79 to 90.19]
  2 Months | 77.95 [70.42 to 83.79] | 75.69 [67.92 to 81.83]
  6 Months | 58.38 [50.03 to 65.82] | 49.42 [40.89 to 57.37]
  12 Months | 49.27 [40.96 to 57.05] | 42.71 [34.39 to 50.75]
  18 Months | 42.94 [34.82 to 50.79] | 37.97 [29.86 to 46.03]
  24 Months | 38.65 [30.50 to 46.72] | 35.55 [27.57 to 43.59]

7. Secondary Outcome: Kaplan Meier Estimates of Probability of Event-free Survival (EFS) by Time Interval
Description: Event-free survival was defined as the time from the date of randomization to the date of hematologic disease relapse/progression, graft failure, or death due to any cause. If a patient was not known to have any event, then EFS was censored at the latest date the patient was known to be alive (on or before the cut-off date). Results are based on Kaplan Meier (KM) estimates.
Time Frame: 1, 2, 6, 12, 18 & 24 months
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 154 | 155
Percentage of participants
  1 Month | 89.38 [83.24 to 93.35] | 82.83 [75.81 to 87.97]
  2 Months | 74.60 [66.82 to 80.82] | 71.72 [63.71 to 78.26]
  6 Months | 53.68 [45.34 to 61.30] | 44.14 [35.82 to 52.13]
  12 Months | 44.53 [36.36 to 52.36] | 39.98 [30.90 to 46.96]
  18 Months | 40.29 [32.30 to 48.12] | 35.09 [27.23 to 43.04]
  24 Months | 34.98 [27.01 to 43.04] | 32.38 [24.61 to 40.37]

8. Secondary Outcome: Cumulative Incidence Rate of Failure-Free Survival (FFS)
Description: FFS was defined as the time from the date of randomization to date of hematologic disease relapse/progression, non-relapse mortality, or addition of new systemic aGvHD treatment.
  Probability of FFS with 95% CIs are presented for each treatment group, accounting for onset of chronic GvHD as the competing risk.
Time Frame: 1, 2, 6, 12, 18, & 24 Months
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Cumulative probability of FFS
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 154 | 155
Cumulative probability of FFS
  1 Month | 17.92 [12.26 to 24.46] | 49.13 [40.94 to 56.80]
  2 Months | 35.39 [27.79 to 43.07] | 61.32 [53.00 to 68.61]
  6 Months | 53.67 [45.28 to 61.34] | 80.17 [72.52 to 85.89]
  12 Months | 58.64 [50.18 to 66.16] | 80.91 [73.32 to 86.54]
  18 Months | 59.35 [50.88 to 66.84] | 80.91 [73.32 to 86.54]
  24 Months | 61.48 [53.01 to 68.88] | 81.66 [74.12 to 87.19]

9. Secondary Outcome: Cumulative Probability of Non Relapse Mortality (NRM)
Description: NRM was defined as the time from date of randomization to date of death not preceded by hematologic disease relapse/progression. Hematologic disease relapse/progression was considered a competing risk for NRM with the date of hematologic disease relapse/progression being the earlier of documented hematologic disease relapse/progression or institution of therapy to treat potential hematologic disease relapse/progression. If a patient was not known to have died or to have relapsed/progressed, then NRM was censored at the latest date the patient was known to be alive (on or before the cut-off date). Data is provided based on cumulative probability of hematologic disease relapse/progression.
Time Frame: 1, 2, 6, 12, 18 & 24 months
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Number (95% Confidence Interval); unit: Cumulative probability of NRM
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 154 | 155
Cumulative probability of NRM
  1 Month | 9.96 [5.83 to 15.39] | 14.52 [9.45 to 20.64]
  2 Months | 20.71 [14.61 to 27.54] | 23.54 [17.04 to 30.65]
  6 Months | 37.59 [29.81 to 45.33] | 42.42 [34.18 to 50.41]
  12 Months | 43.91 [35.75 to 51.77] | 46.11 [37.68 to 54.12]
  18 Months | 46.03 [37.77 to 53.89] | 49.21 [40.63 to 57.22]
  24 Months | 49.53 [40.91 to 57.55] | 49.99 [41.38 to 57.99]

10. Secondary Outcome: Cumulative Probability of Malignancy Relapse/Progression (MR)
Description: MR was defined as the time from date of randomization to hematologic malignancy relapse/progression. Deaths not preceded by hematologic malignancy relapse/progression were considered competing risks. If a patient was not known to have event or competing risks, then MR was censored at the latest date the patient was known to be alive (on or before the cut-off date). Calculated for patients with underlying hematologic malignant disease.
Time Frame: 1, 2, 6, 12 , 18 & 24 months
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization. Calculated for patients with underlying hematologic malignant disease.
Measure: Number (95% Confidence Interval); unit: Cumulative probability of MR
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 147 | 147
Cumulative probability of MR
  1 Month | 0.69 [0.06 to 3.51] | 2.80 [0.92 to 6.54]
  2 Months | 4.21 [1.73 to 8.46] | 4.29 [1.75 to 8.60]
  6 Months | 8.46 [4.60 to 13.79] | 13.49 [8.32 to 19.91]
  12 Months | 10.68 [6.24 to 16.47] | 15.06 [9.56 to 21.71]
  18 Months | 12.91 [7.96 to 19.09] | 16.72 [10.89 to 23.64]
  24 Months | 14.75 [9.32 to 21.37] | 18.81 [12.46 to 26.17]

11. Secondary Outcome: Cumulative Probability of Chronic Graft Versus Host Disease (cGvHD)
Description: Incidence of cGvHD was the time from date of randomization to onset of cGvHD is the diagnosis of any cGvHD including mild, moderate, severe. Deaths without prior onset of cGvHD and hematologic disease relapse/progression were competing risks. If a patient was not known to have event or competing risks, then the incidence of cGvHD was censored at the latest date the patient was known to be alive (on or before the cut-off date).
Time Frame: 1, 2, 6, 12, 18 & 24 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Cumulative probability of cGvHD
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 154 | 155
Cumulative probability of cGvHD
  1 Month | 0 [NA to NA] — N/A: 95% CI could not be achieved as there was no incidence of cGvHD | 1.33 [0.26 to 4.34]
  2 Months | 1.34 [0.26 to 4.39] | 2.03 [0.55 to 5.41]
  6 Months | 15.60 [10.26 to 21.96] | 12.19 [7.40 to 18.25]
  12 Months | 29.66 [22.41 to 37.25] | 20.24 [13.98 to 27.34]
  18 Months | 32.48 [24.96 to 40.20] | 23.36 [16.62 to 30.76]
  24 Months | 36.00 [28.20 to 43.84] | 24.95 [18.00 to 32.50]

12. Secondary Outcome: Exposure-efficacy Relationship of Ruxolitinib in Corticosteroid Refractory aGvHD: PK-Overall Response Rate
Description: Exposure-efficacy relationship of ruxolitinib in terms of concentration-effect and dose-effect.
  ORR was defined as the percentage of participants with a best overall response defined as complete response (CR) or partial response (PR) as assessed by local investigators. CR was defined as a score of 0 for the Acute Graft vs. Host Disease (aGvHD) grading in all evaluable organs that indicates complete resolution of all signs and symptoms of aGvHD in all evaluable organs without administration of additional systemic therapies for any earlier progression, mixed response or non-response of aGvHD.
  PR was defined as improvement of 1 stage in 1 or more organs involved with aGvHD signs or symptoms without progression in other organs or sites without administration of additional systemic therapies for an earlier progression, mixed response or non-response of aGvHD.
Time Frame: Day 28
Population: PK-Efficacy Set: All patients randomized to ruxolitinib treatment arm, who received at least one dose of ruxolitinib, who have post-baseline efficacy data (at least one efficacy parameter) and for whom popPK predictions are available (at least one popPK predicted AUC0-12h).
Measure: Number; unit: Percentage of participants
Arm/Group | Ruxolitinib (RUX)
Number analyzed (Participants) | 118
Percentage of participants | 82.2

13. Secondary Outcome: Exposure-efficacy Relationship of Ruxolitinib in Corticosteroid Refractory aGvHD: PK- Durable Overall Response Rate (DORR)
Description: Exposure-efficacy relationship of ruxolitinib in terms of concentration-effect and dose-effect.
  DORR is the percentage of all participants in each arm who achieved a complete response (CR) or partial response (PR) at Day 28 (primary endpoint) AND maintained a CR or PR at Day 56.
  CR was defined as a score of 0 for the aGvHD grading in all evaluable organs that indicates complete resolution of all signs and symptoms of aGvHD in all evaluable organs without administration of additional systemic therapies for any earlier progression, mixed response or non-response of aGvHD.
  PR was defined as improvement of 1 stage in 1 or more organs involved with aGvHD signs or symptoms without progression in other organs or sites without administration of additional systemic therapies for an earlier progression, mixed response or non-response of aGvHD.
Time Frame: Day 56
Population: PK-Efficacy Set: PK-Efficacy Set: All patients randomized to ruxolitinib treatment arm, who received at least one dose of ruxolitinib, who have post-baseline efficacy data (at least one efficacy parameter) and for whom popPK predictions are available (at least one popPK predicted AUC0-12h).
Measure: Number; unit: Percentage of participants
Arm/Group | Ruxolitinib (RUX)
Number analyzed (Participants) | 67
Percentage of participants | 91.0

14. Secondary Outcome: Exposure-efficacy Relationship of Ruxolitinib in Corticosteroid Refractory aGvHD: PK-Overall Survival
Description: Exposure-efficacy relationship of ruxolitinib in terms of concentration-effect and dose-effect. This represents the percentage of Ruxolitinib-exposed participants dead at 24 months.
  Overall survival (OS) was defined as the time from the date of randomization to date of death due to any cause. If a patient was not known to have died, then OS was censored at the latest date the patient was known to be alive (on or before the cut-off date).the date of death due to any cause.
Time Frame: up to 24 months
Population: as for outcome 13
Measure: Number; unit: Percentage of participants
Arm/Group | Ruxolitinib (RUX)
Number analyzed (Participants) | 150
Percentage of participants | 53.3

15. Secondary Outcome: Best Overall Response Rate (BOR)
Description: Percentage of participants who achieved overall response (OR) (CR+PR) at any time point up to and including Day 28 and before the start of additional systemic therapy for aGvHD.
  CR was defined as a score of 0 for the Acute Graft vs. Host Disease (aGvHD) grading in all evaluable organs that indicates complete resolution of all signs and symptoms of aGvHD in all evaluable organs without administration of additional systemic therapies for any earlier progression, mixed response or non-response of aGvHD.
  PR was defined as improvement of 1 stage in 1 or more organs involved with aGvHD signs or symptoms without progression in other organs or sites without administration of additional systemic therapies for an earlier progression, mixed response or non-response of aGvHD.
Time Frame: up to Day 28
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization. These were participants whose overall response was complete response (CR) or partial response (PR).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 154 | 155
Percentage of participants | 81.8 [74.8 to 87.6] | 60.6 [52.5 to 68.4]
Statistical Analysis 1: Comparison: Ruxolitinib (RUX) vs Best Available Therapy (BAT); Test type: Superiority; p < .0001, Stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.07, 95% CI 2-sided [1.80 to 5.25]

16. Secondary Outcome: Patient Reported Outcomes (PROs): Change From Baseline in Functional Assessment of Cancer Therapy-Bone Marrow Transplantation (FACT-BMT) Total Score
Description: The Functional assessment of Cancer Therapy - Bone Marrow Transplant (FACT-BMT) is a 50-item self-report questionnaire that measures the effect of a therapy on domains including physical, functional, social/family and emotional well-being, together with additional concerns relevant for bone marrow transplantation patients. Patients indicated their response on a scale of 0 to 4 on each statement, with 0 indicating worst score and 4 the best score. All individual scores were combined to calculate the total score. Total score was reported with score range: 0-148 which was calculated as the sum of all unweighted subscale scores. The higher the total score the better the result. Descriptive statistics and change from baseline were calculated in total score at each scheduled assessment time point.
Time Frame: Baseline, Week 24
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 154 | 155
scores on a scale
  Baseline: number analyzed (Participants) | 106 | 94
  Baseline | 89.00 [41.0 to 138.0] | 81.00 [29.0 to 129.0]
  Week (W) 24: number analyzed (Participants) | 36 | 13
  Week (W) 24 | 108.50 [67.0 to 139.0] | 86.00 [21.0 to 124.0]
  Change from Baseline to W24: number analyzed (Participants) | 29 | 12
  Change from Baseline to W24 | 9.00 [-40.0 to 44.0] | 4.50 [-29.0 to 41.0]

17. Secondary Outcome: Patient Reported Outcomes (PROs): Change From Baseline in EuroQol-5D-5L UK Score
Description: The EQ-5D descriptive classification consists of five dimensions of health: mobility, self-care, usual activities, anxiety/depression and pain/discomfort. Patients are requested to select the statement which best describes their condition on that day for each dimension. For overall health that day, the EuroQoL-5D-5L scale is numbered from 0 to 100, with 100 being the best health you can imagine and 0 being the worst health you can imagine. Descriptive statistics (mean, standard deviation, median, Q1, Q3, minimum, and maximum) were calculated based on the scored scales at each scheduled assessment time point. In order to measure Quality-of-Life (QoL) among aGvHD patients, and potential changes over time, change from baseline in EuroQol-5D-5L scores at the time of each assessment were also calculated. Missing items data in a scale will be handled based on each instrument manual. No imputation will be applied if the total or subscale scores are missing at a visit.
Time Frame: Baseline, Week 24
Population: The Full Analysis Set (FAS) comprised all patients to whom study treatment was assigned by randomization.
Measure: Median (Full Range); unit: scores on a scale
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT)
Number analyzed (Participants) | 154 | 155
scores on a scale
  Baseline: number analyzed (Participants) | 122 | 118
  Baseline | 0.60 [-0.6 to 1.0] | 0.54 [-0.6 to 1.0]
  W24: number analyzed (Participants) | 36 | 14
  W24 | 0.78 [0.4 to 1.0] | 0.68 [-0.1 to 1.0]
  Change from Baseline to W24: number analyzed (Participants) | 32 | 12
  Change from Baseline to W24 | 0.12 [-0.3 to 1.1] | 0.12 [-0.2 to 0.3]

18. Secondary Outcome: Pharmacokinetic (PK) Parameter: Area Under the Curve (AUC) (AUCinf, AUClast, AUCtau) of Ruxolitinib
Description: AUClast: The AUC from time zero to the last measurable concentration sampling time (tlast) (mass x time x volume-1) AUCinf: The AUC from time zero to infinity (mass x time x volume-1) AUCtau: The AUC calculated to the end of a dosing interval (tau) at steady-state (amount x time x volume-1).
  Plasma samples for PK was taken at Day 1 (start of treatment), at Day 7 (week 1) to characterize the PK after first dose, and at steady state by non-compartmental analysis.
  The plasma samples from all patients was assayed for ruxolitinib concentrations using validated liquid chromatography-tandem mass spectrometry method (LC-MS/MS).
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 4, 6, 9 hrs post-dose
Population: The Pharmacokinetic Analysis Set (PAS) included all patients who provided at least one evaluable PK concentration. For a concentration to be evaluable, patients were required to: Take a dose of ruxolitinib prior to sampling, Did not vomit within 2 hours after the last dose of ruxolitinib prior to sampling (for pre dose samples) or did not vomit within 2 hours after ruxolitinib dosing (for post dose samples).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Ruxolitinib (RUX)
Number analyzed (Participants) | 26
ng*hr/mL
  Week 1 Day 1 AUCinf: number analyzed (Participants) | 11
  Week 1 Day 1 AUCinf | 529.6 (55.2)
  Week 1 Day 1 AUClast | 522.9 (89.6)
  Week 1 Day 1 AUCtau: number analyzed (Participants) | 20
  Week 1 Day 1 AUCtau | 578.9 (97.5)
  Week 1 Day 7 AUCinf: number analyzed (Participants) | 9
  Week 1 Day 7 AUCinf | 440.9 (91.5)
  Week 1 Day 7 AUClast: number analyzed (Participants) | 22
  Week 1 Day 7 AUClast | 597.3 (73.2)
  Week 1 Day 7 AUCtau: number analyzed (Participants) | 18
  Week 1 Day 7 AUCtau | 651.9 (86.4)

19. Secondary Outcome: Pharmacokinetic (PK) Parameter: Plasma Concentration at Peak (Cmax) of Ruxolitinib
Description: Cmax is the maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration (mass X volume-1).
  Plasma samples for PK was taken at Day 1 (start of treatment), at Day 7 (week 1) to characterize the PK after first dose, and at steady state by non-compartmental analysis.
  The plasma samples from all patients was assayed for ruxolitinib concentrations using validated liquid chromatography-tandem mass spectrometry method (LC-MS/MS).
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 4, 6, 9 hrs post-dose
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ruxolitinib (RUX)
Number analyzed (Participants) | 26
ng/mL
  Week 1 Day 1 | 118 (70.4)
  Week 1 Day 7: number analyzed (Participants) | 22
  Week 1 Day 7 | 129.3 (76.0)

20. Secondary Outcome: Pharmacokinetic (PK) Parameter: CL/F of Ruxolitinib
Description: CL/F is the total body clearance of ruxolitinib from the plasma after a single dose and at steady state.
  Plasma samples for PK was taken at Day 1 (start of treatment), at Day 7 (week 1) to characterize the PK after first dose, and at steady state by non-compartmental analysis.
  The plasma samples from all patients was assayed for Ruxolitinib concentrations using validated liquid chromatography-tandem mass spectrometry method (LC-MS/MS).
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 4, 6, 9 hrs post-dose
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Ruxolitinib (RUX)
Number analyzed (Participants) | 11
L/hr
  Week 1 Day 1 CL/F | 18.88 (55.2)
  Week 1 Day 7 CL/F: number analyzed (Participants) | 9
  Week 1 Day 7 CL/F | 23.31 (89.4)

21. Secondary Outcome: Pharmacokinetic (PK) Parameter: VzF of Ruxolitinib
Description: VzF is the apparent volume of distribution during terminal phase after a single dose and at steady state.
  Plasma samples for PK was taken at Day 1 (start of treatment), at Day 7 (week 1) to characterize the PK after first dose, and at steady state by non-compartmental analysis.
  The plasma samples from all patients will be assayed for ruxolitinib concentrations using validated liquid chromatography-tandem mass spectrometry method (LC-MS/MS).
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 4, 6, 9 hrs post-dose
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Ruxolitinib (RUX)
Number analyzed (Participants) | 11
Liters (L)
  Week 1 Day 1 | 52.57 (46.4)
  Week 1 Day 7: number analyzed (Participants) | 9
  Week 1 Day 7 | 66.76 (71.6)

22. Secondary Outcome: Pharmacokinetic (PK) Parameter: Lambda_z of Ruxolitinib
Description: Lambda_z is the smallest (slowest) disposition (hybrid) rate constant (hr-1) may also be used for terminal elimination rate constant (hr-1).
  Plasma samples for PK was taken at Day 1 (start of treatment), at Day 7 (week 1) to characterize the PK after first dose, and at steady state by non-compartmental analysis.
  The plasma samples from all patients will be assayed for ruxolitinib concentrations using validated liquid chromatography-tandem mass spectrometry method (LC-MS/MS).
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 4, 6, 9 hrs post-dose
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/hr
Arm/Group | Ruxolitinib (RUX)
Number analyzed (Participants) | 11
1/hr
  Week 1 Day 1 | 0.3592 (34.2)
  Week 1 Day 7: number analyzed (Participants) | 9
  Week 1 Day 7 | 0.3492 (31.0)

23. Secondary Outcome: Pharmacokinetic (PK) Parameter: T1/2 of Ruxolitinib
Description: T1/2 is the elimination half-life associated with the terminal slope of a semi logarithmic concentration-time curve (hr).
  Plasma samples for PK was taken at Day 1 (start of treatment), at Day 7 (week 1) to characterize the PK after first dose, and at steady state by non-compartmental analysis.
  The plasma samples from all patients will be assayed for ruxolitinib concentrations using validated liquid chromatography-tandem mass spectrometry method (LC-MS/MS).
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 4, 6, 9 hrs post-dose
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (hr)
Arm/Group | Ruxolitinib (RUX)
Number analyzed (Participants) | 11
hour (hr)
  Week 1 Day 1 | 1.93 (34.2)
  Week 1 Day 7: number analyzed (Participants) | 9
  Week 1 Day 7 | 1.985 (31.0)

24. Secondary Outcome: Pharmacokinetic (PK) Parameter: Tmax of Ruxolitinib
Description: Tmax is the time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after single dose and repeated dose administration (hr).
  Plasma samples for PK was taken at Day 1 (start of treatment), at Day 7 (week 1) to characterize the PK after first dose, and at steady state by non-compartmental analysis.
  The plasma samples from all patients will be assayed for ruxolitinib concentrations using validated liquid chromatography-tandem mass spectrometry method (LC-MS/MS).
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 4, 6, 9 hrs post-dose
Population: as for outcome 18
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Ruxolitinib (RUX)
Number analyzed (Participants) | 26
hour (hr)
  Week 1 Day 1 | 1.767 [0.5167 to 8.917]
  Week 1 Day 7: number analyzed (Participants) | 22
  Week 1 Day 7 | 1.542 [0.5 to 4.083]

25. Secondary Outcome: Pharmacokinetic (PK) Parameter: Racc of Ruxolitinib
Description: Racc is the accumulation ratio (AUC at steady state/AUC Day 1). Plasma samples for PK was taken at Day 1 (start of treatment), at Day 7 (week 1) to characterize the PK after first dose, and at steady state by non-compartmental analysis.
  The plasma samples from all patients was be assayed for ruxolitinib concentrations using validated liquid chromatography-tandem mass spectrometry method (LC-MS/MS).
Time Frame: pre-dose, 0.5, 1, 1.5, 2, 4, 6, 9 hrs post-dose
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Ruxolitinib (RUX)
Number analyzed (Participants) | 26
ratio | 1.145 (27.2)

26. Secondary Outcome: Pharmacokinetic (PK) Parameter: Ctrough of Ruxolitinib
Description: Minimum concentration (Ctrough) of ruxolitinib and at steady state in corticosteroid refractory acute GVHD patients.
  Plasma samples for PK was taken at Day 1 (start of treatment), at Day 7 (week 1) to characterize the PK after first dose, and at steady state by non-compartmental analysis.
  The plasma samples from all patients will be assayed for ruxolitinib concentrations using validated liquid chromatography-tandem mass spectrometry method (LC-MS/MS)
Time Frame: pre-dose
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/ml
Arm/Group | Ruxolitinib (RUX)
Number analyzed (Participants) | 152
ng/ml | 17.22 (187.1)

27. Post Hoc Outcome: All Collected Deaths
Description: On treatment deaths were collected from the start of treatment up to 30 days after study drug discontinuation, for a maximum duration of 708 days (treatment duration ranged from 6.0 to 678.0) for the RUX arm and 218 days (treatment duration ranged from 1.0 to 188.0 days) for the BAT arm.
  Deaths post treatment survival follow up were collected after the on- treatment period, up to approx. 48 months. Patients who didn't die during the on-treatment period and had not stopped study participation at the time of data cut-off (end of study) were censored.
Time Frame: approx. 708 days (AEs), up to approx. 48 months (deaths)
Population: Clinical Database Population: all randomized patients
Measure: Number; unit: Participants
Groups:
- Cross-Over: These were patients randomized to BAT who were eligible to cross over to Ruxolitinib between Day 28 and Week 24.
Arm/Group | Ruxolitinib (RUX) | Best Available Therapy (BAT) | Cross-Over
Number analyzed (Participants) | 152 | 150 | 49
Participants
  Total Deaths | 89 | 89 | 29
  Deaths on-treatment | 43 | 36 | 19

ADVERSE EVENTS:
Time Frame: On treatment deaths were collected from the start of treatment up to 30 days after study drug discontinuation, for a maximum duration of 708 days (treatment duration ranged from 6.0 to 678.0) for the RUX arm and 218 days (treatment duration ranged from 1.0 to 188.0 days) for the BAT arm. Deaths occurred from Randomization till end of the study, up to approx. 48 months.
Description: Adverse Event (AE): Any sign or symptom that occurs during treatment plus 30 days post treatment.
Arm/Group | Ruxolitinib (Rux) | Best Available Therapy (BAT) | Cross-Over
All-Cause Mortality (participants affected / at risk) | 89/152 | 89/150 | 29/49
Serious Adverse Events (participants affected / at risk) | 101/152 | 80/150 | 38/49
Other Adverse Events (participants affected / at risk) | 144/152 | 136/150 | 43/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (Rux) (N=152) | Best Available Therapy (BAT) (N=150) | Cross-Over (N=49)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 0
Haemolysis (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Myelosuppression (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 2
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 2 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 3 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 2
Ileal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Ileal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 2
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Condition aggravated (General disorders) | 1 | 0 | 1
Disease recurrence (General disorders) | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 3 | 0
Pyrexia (General disorders) | 10 | 6 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Acute graft versus host disease (Immune system disorders) | 2 | 2 | 0
Acute graft versus host disease in intestine (Immune system disorders) | 0 | 2 | 0
Allergy to immunoglobulin therapy (Immune system disorders) | 0 | 1 | 0
Graft versus host disease (Immune system disorders) | 0 | 3 | 1
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 1 | 0 | 0
Serum sickness (Immune system disorders) | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0
Adenovirus infection (Infections and infestations) | 0 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 4 | 1
Bacterial disease carrier (Infections and infestations) | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 1
Cerebral aspergillosis (Infections and infestations) | 1 | 0 | 0
Clostridial sepsis (Infections and infestations) | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Cystitis viral (Infections and infestations) | 2 | 0 | 0
Cytomegalovirus colitis (Infections and infestations) | 3 | 0 | 0
Cytomegalovirus enteritis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 3 | 2 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 3 | 6 | 2
Device related infection (Infections and infestations) | 1 | 1 | 1
Encephalitis (Infections and infestations) | 0 | 0 | 1
Encephalitis viral (Infections and infestations) | 0 | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 0 | 0 | 1
Enterobacter sepsis (Infections and infestations) | 1 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Enterococcal infection (Infections and infestations) | 1 | 0 | 0
Escherichia infection (Infections and infestations) | 2 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 1 | 0
Fungal sepsis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 1 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 2 | 1 | 0
Intestinal sepsis (Infections and infestations) | 0 | 1 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection fungal (Infections and infestations) | 0 | 0 | 1
Meningitis enterococcal (Infections and infestations) | 0 | 0 | 1
Mucormycosis (Infections and infestations) | 2 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 2 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 7 | 8 | 2
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 2 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1 | 1
Pseudomonal sepsis (Infections and infestations) | 3 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 12 | 10 | 7
Septic shock (Infections and infestations) | 10 | 8 | 3
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 2 | 1 | 0
Systemic candida (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection viral (Infections and infestations) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0 | 0
Viral infection (Infections and infestations) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Graft loss (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Transplantation complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bacterial test positive (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 3 | 0 | 0
Cytomegalovirus test positive (Investigations) | 0 | 0 | 1
General physical condition abnormal (Investigations) | 2 | 0 | 0
Influenza B virus test positive (Investigations) | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 1
Oxygen saturation decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 3 | 1
Transaminases increased (Investigations) | 0 | 0 | 1
White blood cell count decreased (Investigations) | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Acute erythroid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
Chorea (Nervous system disorders) | 0 | 0 | 1
Coma (Nervous system disorders) | 1 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 2 | 2 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Mononeuropathy (Nervous system disorders) | 0 | 1 | 0
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 1 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1
Stupor (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 3 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 5 | 2
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 3 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 1 | 0
Perineal ulceration (Reproductive system and breast disorders) | 0 | 1 | 0
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Idiopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 6
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Embolism (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1
Microangiopathy (Vascular disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib (Rux) (N=152) | Best Available Therapy (BAT) (N=150) | Cross-Over (N=49)
Anaemia (Blood and lymphatic system disorders) | 61 | 47 | 16
Leukopenia (Blood and lymphatic system disorders) | 14 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 36 | 19 | 10
Thrombocytopenia (Blood and lymphatic system disorders) | 56 | 30 | 14
Tachycardia (Cardiac disorders) | 3 | 9 | 2
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 20 | 11 | 4
Constipation (Gastrointestinal disorders) | 9 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 18 | 20 | 4
Nausea (Gastrointestinal disorders) | 30 | 16 | 3
Stomatitis (Gastrointestinal disorders) | 6 | 5 | 3
Vomiting (Gastrointestinal disorders) | 25 | 16 | 5
Fatigue (General disorders) | 11 | 6 | 3
Generalised oedema (General disorders) | 5 | 8 | 0
Oedema peripheral (General disorders) | 37 | 32 | 5
Pyrexia (General disorders) | 29 | 21 | 9
Hypogammaglobulinaemia (Immune system disorders) | 14 | 7 | 3
Cytomegalovirus infection (Infections and infestations) | 11 | 9 | 1
Cytomegalovirus infection reactivation (Infections and infestations) | 38 | 30 | 8
Device related infection (Infections and infestations) | 13 | 5 | 1
Epstein-Barr virus infection reactivation (Infections and infestations) | 8 | 6 | 1
Pneumonia (Infections and infestations) | 10 | 6 | 3
Sepsis (Infections and infestations) | 5 | 9 | 3
Urinary tract infection (Infections and infestations) | 15 | 9 | 1
Fall (Injury, poisoning and procedural complications) | 12 | 3 | 2
Alanine aminotransferase increased (Investigations) | 16 | 11 | 2
Aspartate aminotransferase increased (Investigations) | 9 | 9 | 1
Blood bilirubin increased (Investigations) | 7 | 15 | 3
Blood creatinine increased (Investigations) | 8 | 10 | 3
C-reactive protein increased (Investigations) | 4 | 5 | 3
Gamma-glutamyltransferase increased (Investigations) | 14 | 12 | 2
Neutrophil count decreased (Investigations) | 19 | 16 | 4
Platelet count decreased (Investigations) | 31 | 24 | 6
Weight decreased (Investigations) | 7 | 5 | 3
White blood cell count decreased (Investigations) | 21 | 16 | 2
Decreased appetite (Metabolism and nutrition disorders) | 7 | 8 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 15 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 9 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 9 | 4 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18 | 20 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 16 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 34 | 28 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 23 | 23 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 6 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 15 | 15 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7 | 4
Myopathy (Musculoskeletal and connective tissue disorders) | 7 | 9 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 10 | 0
Headache (Nervous system disorders) | 13 | 5 | 2
Tremor (Nervous system disorders) | 6 | 5 | 3
Depression (Psychiatric disorders) | 9 | 4 | 1
Insomnia (Psychiatric disorders) | 9 | 8 | 2
Acute kidney injury (Renal and urinary disorders) | 18 | 7 | 2
Dysuria (Renal and urinary disorders) | 8 | 6 | 0
Haematuria (Renal and urinary disorders) | 12 | 6 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 12 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 8 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Hypertension (Vascular disorders) | 21 | 18 | 6
Hypotension (Vascular disorders) | 15 | 10 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Study Protocol (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT02913261/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT02913261/SAP_001.pdf